CLINICAL TRIAL: NCT03355755
Title: Exoskeleton Treatment of Deconditioning Due to Limited Ambulation Caused by Illness or Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ekso Bionics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 107159
Record Dates: First submitted 2017-11-03; First posted 2017-11-28 (Actual); Results first posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Debility Due to Disease

STUDY DESIGN:
Intervention Model Description: Single-arm safety and feasibility study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Interventional Group (Experimental): All participants will be included in the interventional group. Intervention will consist of walking exercise using the EksoGT exoskeleton for supported walking, running SmartAssist software.
  Interventions: Device: EksoGT with SmartAssist software

INTERVENTIONS:
Device: EksoGT with SmartAssist software — Intervention will consist of exercise using the EksoGT exoskeleton for supported walking. The EksoGT is a powered motorized orthosis intended to enable individuals who are experiencing muscular or neurological conditions affecting their lower extremities to perform ambulatory functions such as gait training.

SUMMARY:
A safety and feasibility study of robotic exoskeleton training in deconditioned patients residing in a healthcare facility.

DETAILED DESCRIPTION:
Patients who are hospitalized for several weeks or months are at a higher risk of decline in physical condition and are also at a higher risk of rehospitalization within 30 days of discharge. A program incorporating robotic exoskeleton training may provide sufficient physical support and challenge for patients to maintain a higher level of physical condition than if they did not undergo exoskeleton training. The investigators aim to demonstrate that EksoGT robotic exoskeleton training can be performed safely with patients who have been hospitalized and are at risk of experiencing a further decline in their physical condition.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of "deconditioned", defined as the loss of muscle tone and endurance due to chronic disease, immobility, or loss of function.
2. Adults 18 years and older (or as specified by state law).
3. Admitted into a hospital, long-term care facility, skilled nursing facility, or similar.
4. Sufficient upper extremity strength to use a front wheeled walker by manual muscle testing (minimum triceps strength bilaterally of 3/5, shoulder abduction and flexion/extension 4/5).
5. Screened and cleared by a physician for full weight-bearing exercise training.
6. Weigh 220 pounds (100kg) or less.
7. Between approximately 5'0" and 6'4" tall.
8. Standing hip width of approximately 18" or less.
9. Have near normal range of motion in hips, knees and ankles.

Exclusion Criteria:

1. Currently involved in another intervention study.
2. Transferred to the intensive care unit or isolation-room stay.
3. Currently on a ventilator or extracorporeal membrane oxygenation (ECMO) machine.
4. Currently have a ventricular assist device (VAD) or an automatic implantable cardioverter-defibrillator (AICD).
5. Advanced heart failure - ejection fraction of < 20%.
6. Documented cardiovascular risk from exercise.
7. Resting heart rate <50 bpm or >120 bpm.
8. Uncontrolled or new (within 24 hours) arrythmias.
9. Resting blood pressure below 90/70 or above 160/100.
10. Oxygen saturation (O2 sat) < 90% during rest.
11. Uncontrolled or severe orthostatic hypotension that limits standing tolerance.
12. Cardiac ischemia within 24 hours.
13. Unresolved or new (within 24 hours) deep vein thrombosis.
14. Concurrent severe neurological pathology/disease or stroke within 72 hours.
15. Open skin ulcerations on any body surfaces in contact with exoskeleton.
16. Acute fracture
17. Osteoporosis
18. Active heterotrophic ossification (HO) of the lower extremity, hip dysplasia, or hip/knee axis abnormalities.
19. Current chemotherapy
20. Inability to speak or understand the English language.
21. Inability to cooperate in tests/exercises.
22. Hip flexion contracture greater than ~17°.
23. Knee flexion contracture greater than 12°.
24. Unable to achieve neutral ankle dorsiflexion with passive stretch (neutral with max 12° knee flexion).
25. Cognitive impairments - unable to follow 2 step commands or to communicate pain or to stop session.
26. Pregnancy
27. Any reason the physician may deem as harmful to the participant to enroll or continue in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Gaylord Specialty Healthcare, Wallingford, Connecticut
  - Marianjoy Rehabilitation Hospital, Wheaton, Illinois
  - Quality Living, Inc, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomas JI, Lane JV. A pilot study to explore the predictive validity of 4 measures of falls risk in frail elderly patients. Arch Phys Med Rehabil. 2005 Aug;86(8):1636-40. doi: 10.1016/j.apmr.2005.03.004. PMID 16084819
- [Background] Hoyer EH, Needham DM, Miller J, Deutschendorf A, Friedman M, Brotman DJ. Functional status impairment is associated with unplanned readmissions. Arch Phys Med Rehabil. 2013 Oct;94(10):1951-8. doi: 10.1016/j.apmr.2013.05.028. Epub 2013 Jun 26. PMID 23810355
- [Background] Hoyer EH, Needham DM, Atanelov L, Knox B, Friedman M, Brotman DJ. Association of impaired functional status at hospital discharge and subsequent rehospitalization. J Hosp Med. 2014 May;9(5):277-82. doi: 10.1002/jhm.2152. Epub 2014 Feb 26. PMID 24616216
- [Background] Hoyer EH, Brotman DJ, Chan KS, Needham DM. Barriers to early mobility of hospitalized general medicine patients: survey development and results. Am J Phys Med Rehabil. 2015 Apr;94(4):304-12. doi: 10.1097/PHM.0000000000000185. PMID 25133615
- [Background] Hoyer EH, Friedman M, Lavezza A, Wagner-Kosmakos K, Lewis-Cherry R, Skolnik JL, Byers SP, Atanelov L, Colantuoni E, Brotman DJ, Needham DM. Promoting mobility and reducing length of stay in hospitalized general medicine patients: A quality-improvement project. J Hosp Med. 2016 May;11(5):341-7. doi: 10.1002/jhm.2546. Epub 2016 Feb 5. PMID 26849277

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One arm study.
Period: Overall Study
Arm/Group | Interventional Group
Started | 15
Completed | 13
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Interventional Group
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.87 (19.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 15
Days since diagnosis [Mean (Standard Deviation); unit: days] — From study initiation, how many days prior had patient been diagnosed with deconditioning Population: One participants date of diagnosis was unknown and not analyzed
  days
    number analyzed (Participants) | 14
    (all) | 93.62 (75.54)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience an Adverse Event During Time of Treatment
Description: The primary endpoint is safety defined as the number of participants experiencing an adverse event per overall during the study period.
Time Frame: 2 weeks
Population: 2 participants did not complete study protocol due to early discharge from hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Group
Number analyzed (Participants) | 13
Participants | 5

2. Secondary Outcome: Number of Participants Who Experience an Adverse Event During Time of Treatment That Was Deemed "Definitely Device Related"
Description: Count of number of participants who experienced any adverse event that was rated as definitely related to treatment with the Ekso device.
Time Frame: 2 weeks
Population: 2 participants did not complete study protocol due to early discharge from hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Group
Number analyzed (Participants) | 13
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events were taken through the duration of the study (completing 5 sessions in exoskeleton) which took, on average, 12 days to complete.
Arm/Group | Interventional Group
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 5/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional Group (N=13)
Fall (Injury, poisoning and procedural complications) | 3 (3) — Three participants experienced single fall in which no injuries were documented and no medical treatment was necessary
skin tear and pressure sores (Skin and subcutaneous tissue disorders) | 2 (2) — one participant experienced a consistent pressure ulcer session 1-4. Another participant experienced a minor right posterior thigh skin tear requiring no medical intervention
Spasm (Nervous system disorders) | 1 (1) — One participant experienced an increase in nightime spasm
Swelling and erythema (Skin and subcutaneous tissue disorders) | 1 (1) — One participant experienced a single episode of leg swelling and erythema on anterior shins both categorized as mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT03355755/Prot_001.pdf